CLINICAL TRIAL: NCT04091906
Title: Peripheral Blood Mononuclear Cell Donation Protocol for Tumor Immunotherapy Study of UCAR-T Cells
Brief Title: PBMC Donation in UCAR-T Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JSPH-CTA101-PBMC
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Peripheral Blood Mononuclear Cell Donation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy donor (Experimental)
  Interventions: Device: Peripheral blood mononuclear cell apheresis

INTERVENTIONS:
Device: Peripheral blood mononuclear cell apheresis — Peripheral blood mononuclear cell donation for tumor immunotherapy study of UCAR-T cells

SUMMARY:
Peripheral blood mononuclear cell donation protocol for tumor immunotherapy study of UCAR-T cells

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-40 years, no donation reaction in the past;
2. Weight: male ≥ 50 kg, female ≥ 45 kg, and 18.5 kg/m2 ≤ BMI ≤ 30 kg/m2;
3. Blood pressure:

12.0 Kpa (90 mmHg) ≤ systolic pressure﹤18.7 Kpa (140 mmHg) 8.0 Kpa (60 mmHg) ≤ diastolic pressure﹤12.0 Kpa (90 mmHg) Pulse pressure ≥ 4.0Kpa (30mmHg); 4) Pulse: 60/min to 100/min. Athletes with high endurance ≥ 50/min, with regular rhythm; 5) Temperature: 36.3-37.2℃ (oral temperature); 6) Generally in good condition: no damage to important organs such as heart, lung, liver and kidney; no severe or uncontrolled infection; no history of severe mental disorders; 7) Clinical examination should meet the following criteria:

1. Hemoglobinometry: male ≥ 120g/L; female ≥ 110g/L. If using copper sulfate method: male ≥ 1.0520, female ≥ 1.0510
2. White blood cell (WBC) test: ≥4×109/L
3. Alanine aminotransferase (ALT) ≤40U/L (Rate method), ≤25U/L (Reitman-Frankel method)
4. Hepatitis B virus surface antigen (HBsAg) negative
5. Hepatitis C virus antibody (HCV antibody) negative
6. Human immunodeficiency virus antibody (HIV-1 and HIV-2 antibody) negative
7. Syphilis negative
8. Cytomegalovirus antibody (CMV antibody) negative
9. Epstein-Barr virus antibody (EBV antibody) negative

Exclusion Criteria:

Donors are ineligible to donate PBMC under the following circumstances:

1) Valetudinarian, with frequent dizziness, giddiness, tinnitus, hemophobia, fear of needles, faint, and Meniere's disease; 2) Sexually transmitted diseases (STDs), leprosy, AIDS, and HIV-1, HIV-2, CMV, EBV antibody positive; 3) History of liver diseases, HBsAg positive and HCV antibody positive. 1 year after the clinical cure of hepatitis A, normal ALT test results at 1 month interval for 3 consecutive times; 4) Relapsed allergic diseases, urticaria, bronchial asthma and drug allergies (Donors with simple urticaria who are not in acute attack are eligible to donate PBMC); 5) Pulmonary tuberculosis, renal tuberculosis, lymph node tuberculosis and bone tuberculosis; 6) Cardiovascular disease and history, various heart diseases, hypertension, hypotension, myocarditis and thrombophlebitis; 7) Respiratory diseases (including chronic bronchitis, emphysema, bronchiectasis and pulmonary insufficiency); 8) Digestive system diseases (e.g. severe gastric and duodenal ulcers, chronic gastroenteritis and chronic pancreatitis); 9) Urinary system diseases (e.g. acute and chronic nephritis, chronic urinary system infection, nephrotic syndrome, acute and chronic renal insufficiency, etc.); 10) Various hematological diseases (including anemia, leukemia, polycythemia vera and various hemorrhagic and coagulative diseases); 11) Endocrine diseases or metabolic disorders (e.g. hyperthyroidism, acromegaly, diabetes insipidus, diabetes mellitus, etc.); 12) Organic nervous system diseases or psychoses (e.g. encephalitis, sequelae of brain trauma, epilepsy, schizophrenia, hysteria, severe neurasthenia, etc.); 13) Parasitic diseases and endemic diseases (e.g. kala-azar, schistosomiasis, filariasis, hookworm disease, taeniasis, paragonimiasis, Keshan disease, Kaschin-Beck disease, etc.); 14) Malignancies and benign tumors affecting health; 15) History of haematological malignancies (e.g. leukaemia, lymphoma, myeloma), history of malignancies known to be associated with viraemic conditions (except for carcinoma in situ of the cervix). For other cancers, the donors should have fully recovered with no expectation of recurrence (i.e. cured) and the following conditions apply:

1. for cancers with negligible metastatic potential (e.g. basal cell carcinoma and carcinoma in situ of the cervix), the donors may be accepted immediately following successful removal and cure
2. for all other cancers, at least 5 years should have elapsed since completion of active treatment 16) Undergone resection of stomach, kidney, gallbladder, spleen, lung and other important organs; 17) Exposure to harmful substances or radioactive substances (except for clinical radiology); 18) High-risk groups susceptible to HIV infection, such as drug users, homosexuals and people with multiple sexual partners; 19) Creutzfeldt-Jakob disease (CJD), variant Creutzfeldt disease (vCJD), family history, and treatment with human and animal pituitary-derived substances (e.g. growth hormone, gonadotropin, thyrotropin, etc.). Organ transplantation recipients (including cornea, bone marrow, dura mater) may be exposed to bovine spongiform encephalopathy (BSE) and vCJD; 20) Chronic skin diseases, especially infectious, allergic and inflammatory systemic skin diseases (e.g. favus, generalized eczema, systemic psoriasis, etc.); 21) Autoimmune diseases and collagenosis (e.g. systemic lupus erythematosus, dermatomyositis, scleroderma, etc.); 22) Bitten by animals carrying rabies virus; 23) Other diseases or conditions in which donors are ineligible to donate PBMC in the opinion of physicians;

Donors should be deferred for the time being under the following circumstances:

1. Tooth extraction or other minor surgery within half a month;
2. 3 days before or after menstruation, menstrual disorders, pregnancy, less than 6 months after abortion, less than 1 year after delivery and lactation;
3. Less than 1 week after the recovery of cold and acute gastroenteritis, less than 1 month after the cure of acute urinary system infection, and less than half a year after the cure of pneumonia;
4. Donors from high-risk areas of infectious diseases as prescribed by certain infectious diseases and epidemic prevention departments. Less than half a year after the cure of dysentery, less than 1 year after the cure of typhoid fever and brucellosis, history of malaria within 3 years;
5. Within 2 years after blood transfusion treatment;
6. Less than 1 year after tattoo, injuries or contaminated wounds caused by equipment contaminated by blood or tissue fluid;
7. Close contact history with patients with infectious diseases: within the longest incubation period of the disease after the date of contact;
8. Recipients of animal serum products: within 4 weeks after the last injection;
9. Recipients of hepatitis B immunoglobulin (HBIG) injection: within 1 year;

Provisions for PBMC collection after immunization:

1) Asymptomatic donors who have recently received immunization may donate PBMC only after the following period of time: 2 weeks after the last immunization of measles, mumps, yellow fever, poliomyelitis and live attenuated hepatitis A vaccine, 4 weeks after the last immunization of live rubella vaccine and rabies vaccine;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Collect blood samples | Baseline
  Collect blood samples (whole blood and PBMC) from healthy donors for the development and production of UCAR-T cells

SECONDARY OUTCOMES:
Collect blood samples | Baseline
  Collect blood samples (whole blood) for pre-preparation of autologous CAR-T cells, comparation with UCAR-T products, exploration of the differences in cell expansion and function between UCAR-T and autologous CAR-T, and pre-experiments in the development of various test methodologies

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China